CLINICAL TRIAL: NCT00294151
Title: Challenging the Paradigm in Pain Relief for Advanced Breast and Prostate Cancer Patients With Vertebral Metastasis: Vertebral Augmentation With Cement Plus Radiotherapy Versus Radiotherapy. A Randomized, Prospective, Double Blind Pilot Study
Brief Title: Potential Vertebroplasty Use in the Treatment of Vertebral Metastasis From Breast and Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEN#05-015
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2006-01

CONDITIONS: Breast Cancer; Prostate Cancer; Vertebral Metastasis; Pain
Keywords: breast cancer; prostate cancer; vertebral metastasis; vertebroplasty; vertebral metastasis from breast cancer; vertebral metastasis from prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Pain | interventions — Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty

SUMMARY:
The study aims to evaluate if adding vertebroplasty to radiotherapy, in the treatment of spine metastasis from breast and prostate cancer, is preferable to radiotherapy alone. The investigators hypothesize that, by combining vertebral augmentation with cement and radiotherapy, they could achieve an enhancement in pain relief and level of activities, as well as a decrease in the side effects of multiple medications used for pain control.

DETAILED DESCRIPTION:
Included patients presenting with spinal metastasis secondary to breast or prostate cancer are randomized to two groups, intervention and control. Both groups receive standard radiotherapy, which is currently the gold standard of care for such patients. The intervention group will also receive a vertebroplasty [single or multiple level(s)], while the control group will receive a simulated vertebroplasty, where local anesthesia and gentle hand manipulation will be used but the vertebra will not be accessed. The primary outcome is pain relief, though other factors such as quality of life and pain medications will also be evaluated.

There will be an interim analysis after half of the patients have been treated with a follow-up of 3 months. In the analysis, comparisons will be made between the two groups and each patient's individual progress will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between 35 and 75 years old
* Biopsy-proven breast cancer (BC) or prostate cancer (PC)
* Radiographic evidence of spine metastases from the BC or PC in the lumbar and/or mid-low thoracic spine
* Microfractures or compression fractures up to 40% of the original height of the vertebral body in an MRI [magnetic resonance imaging] (reported by an independent radiologist)
* Incidental back pain (Verbal Analog Scale > 5/10) felt to be related to those metastases

Exclusion Criteria:

* Spinal cord compression
* Massive rupture of the posterior wall of the vertebral body (according to blinded radiological report)
* Coagulopathy (International Normalized Ratio [INR] > 1.5, platelets < 80,000)
* Inability to communicate in English, French or Spanish
* Previous radiotherapy to the spine in the area presently affected
* Mental cognitive impairment
* Vertebral metastasis without fracture in the MRI

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
pain relief; score on pain questionnaire | at baseline, 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after

SECONDARY OUTCOMES:
quality of life; score on 2 quality of life questionnaires | at baseline, 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after
pain medication | listed at baseline, 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after
side effects | listed at 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after
cost of medical care | evaluated at baseline, 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after
survival | recorded at 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after
new vertebral fractures | recorded at 1 week, 2 weeks, 4 weeks, 3 months, 6 months, 1 year after

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Asenjo, MD, Principal Investigator — Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Saarto T, Janes R, Tenhunen M, Kouri M. Palliative radiotherapy in the treatment of skeletal metastases. Eur J Pain. 2002;6(5):323-30. doi: 10.1016/s1090-3801(02)00028-9. PMID 12160506
- [Background] Wu JS, Bezjak A, Chow E, Kirkbride P. Primary treatment endpoint following palliative radiotherapy for painful bone metastases: need for a consensus definition? Clin Oncol (R Coll Radiol). 2002 Feb;14(1):70-7. doi: 10.1053/clon.2001.0012. PMID 11899906
- [Background] McQuay HJ. The Cochrane Database of Systematic Reviews 3:---,2003.
- [Background] McLain R. Tumors of the Spine. In Herkowitz H et al. The Spine Philadelphia, WB Saunders Co 1171-1206, 1999.
- [Background] Niv D, Gofeld M, Devor M. Causes of pain in degenerative bone and joint disease: a lesson from vertebroplasty. Pain. 2003 Oct;105(3):387-392. doi: 10.1016/S0304-3959(03)00277-X. PMID 14527699
- [Background] Molloy S, Mathis JM, Belkoff SM. The effect of vertebral body percentage fill on mechanical behavior during percutaneous vertebroplasty. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1549-54. PMID 12865843